CLINICAL TRIAL: NCT02032901
Title: A Phase 3 Evaluation of Daclatasvir and Sofosbuvir in Treatment Naive and Treatment Experienced Subjects With Genotype 3 Chronic Hepatitis C Infection
Brief Title: Phase III Daclatasvir and Sofosbuvir for Genotype 3 Chronic HCV
Acronym: ALLY 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI444-218
Record Dates: First submitted 2014-01-09; First posted 2014-01-10 (Estimated); Results first posted 2015-09-14 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — daclatasvir; Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A1:Daclatasvir + Sofosbuvir in treatment-naive subjects (Experimental): Daclatasvir 60 mg tablet and Sofosbuvir 400 mg tablet orally once daily for 12 weeks
  Interventions: Drug: Daclatasvir; Drug: Sofosbuvir
- A2:Daclatasvir + Sofosbuvir in treatment-experienced subjects (Experimental): Daclatasvir 60 mg tablet and Sofosbuvir 400 mg tablet orally once daily for 12 weeks
  Interventions: Drug: Daclatasvir; Drug: Sofosbuvir

INTERVENTIONS:
Drug: Daclatasvir
  Other Names: BMS-790052
Drug: Sofosbuvir

SUMMARY:
To study the combination of Daclatasvir and Sofosbuvir for the treatment of hepatitis C virus (HCV) Genotype 3 infection

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Key Inclusion Criteria:

* Subjects must be able to understand and agree to comply with the prescribed dosing regimens and procedures, report for regularly scheduled study visits, and reliably communicate with study personnel about adverse events and concomitant medications
* Subjects chronically infected with hepatitis C virus (HCV) genotype 3
* Subjects who are HCV treatment-naive
* Subjects who are HCV treatment-experienced (previous exposure to non-structural 5A inhibitors is prohibited)
* HCV RNA ≥10,000 IU/mL at screening

Key Exclusion Criteria:

* HCV Genotypes other than genotype-3 infection; mixed genotype infections are not permitted
* Liver or any other organ transplant (including hematopoietic stem cell transplants) other than cornea and hair
* Current or known history of cancer (except in situ carcinoma of the cervix or adequately treated basal or squamous cell carcinoma of the skin) within 5 years prior to screening
* Documented or suspected hepatocellular carcinoma, as evidenced by previously obtained imaging studies or liver biopsy (or on a screening imaging study/liver biopsy if this was performed)
* Evidence of decompensated liver disease including, but not limited to, radiologic criteria, a history or presence of ascites, bleeding varices, or hepatic encephalopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (31):
- United States (30):
  - Scripps Clinic, La Jolla, California
  - Peter J Ruane MD Inc, Los Angeles, California
  - National Research Institute, Los Angeles, California
  - Anthony M. Mills MD Inc, Los Angeles, California
  - Huntington Medical Research Institutes, Pasadena, California
  - Precision Research Institute, LLC, San Diego, California
  - Medical Associates Research Group, San Diego, California
  - Quest Clinical Research, San Francisco, California
  - Midland Florida Clinical Research Center, LLC, DeLand, Florida
  - University of Florida Hepatology Research, Gainesville, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Gastrointestinal Specialists Of Georgia, Marietta, Georgia
  - Dupage Medical Group, Downers Grove, Illinois
  - Mercy Medical Center, Inc., Baltimore, Maryland
  - Digestive Disease Associates, P.A., Baltimore, Maryland
  - Kansas City Research Institute, Kansas City, Missouri
  - Southwest Care Center, Santa Fe, New Mexico
  - North Shore University Hospital, Manhasset, New York
  - Premier Medical Group Of The Hudson Valley, Pc, Poughkeepsie, New York
  - Asheville Gastroenterology Associates, PA, Asheville, North Carolina
  - Digestive Health Specialists, PA, Winston-Salem, North Carolina
  - Main Line Gastroenterology Associates Pc, Perkasie, Pennsylvania
  - Center For Liver Diseases, Pittsburgh, Pennsylvania
  - Gastro One, Germantown, Tennessee
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - American Research Corporation, San Antonio, Texas
  - Clinical Research Centers Of America, Murray, Utah
  - Lifetree Clinical Research, Salt Lake City, Utah
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
- Fundacion De Investigacion De Diego, San Juan, Puerto Rico

REFERENCES:
- [Derived] Kowdley KV, Nelson DR, Lalezari JP, Box T, Gitlin N, Poleynard G, Rabinovitz M, Ravendhran N, Sheikh AM, Siddique A, Bhore R, Noviello S, Rana K. On-treatment HCV RNA as a predictor of sustained virological response in HCV genotype 3-infected patients treated with daclatasvir and sofosbuvir. Liver Int. 2016 Nov;36(11):1611-1618. doi: 10.1111/liv.13165. Epub 2016 Jun 16. PMID 27188960
- [Derived] Nelson DR, Cooper JN, Lalezari JP, Lawitz E, Pockros PJ, Gitlin N, Freilich BF, Younes ZH, Harlan W, Ghalib R, Oguchi G, Thuluvath PJ, Ortiz-Lasanta G, Rabinovitz M, Bernstein D, Bennett M, Hawkins T, Ravendhran N, Sheikh AM, Varunok P, Kowdley KV, Hennicken D, McPhee F, Rana K, Hughes EA; ALLY-3 Study Team. All-oral 12-week treatment with daclatasvir plus sofosbuvir in patients with hepatitis C virus genotype 3 infection: ALLY-3 phase III study. Hepatology. 2015 Apr;61(4):1127-35. doi: 10.1002/hep.27726. Epub 2015 Mar 10. PMID 25614962
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 31 sites in 2 countries.
Pre-assignment Details: A total of 173 participants were enrolled in the study. 152 were treated. 21 participants were not treated as they no longer met the study criteria.
Groups:
- Daclatasvir + Sofosbuvir in Treatment-naive Participants: Participants infected with hepatitis C virus (HCV) genotype-3 and not exposed to an interferon formulation or ribavirin or any other HCV-specific direct-acting antiviral therapy, received daclatasvir 60-mg and sofosbuvir 400-mg tablets orally once daily for 12 weeks.
- Daclatasvir + Sofosbuvir in Treatment-experienced Participants: Participants infected with hepatitis C virus (HCV) genotype-3 and previously exposed to an interferon formulation or sofosbuvir /ribavirin or any other anti-HCV agents therapy, received daclatasvir 60-mg tablets and sofosbuvir 400-mg tablets orally once daily for 12 weeks.
Period: Treatment Period (12 Weeks)
Arm/Group | Daclatasvir + Sofosbuvir in Treatment-naive Participants | Daclatasvir + Sofosbuvir in Treatment-experienced Participants
Started | 101 | 51
Completed | 100 | 51
Not Completed | 1 | 0
Not completed — Pregnancy | 1 | 0
Period: Follow-Up Period (24 Weeks)
Arm/Group | Daclatasvir + Sofosbuvir in Treatment-naive Participants | Daclatasvir + Sofosbuvir in Treatment-experienced Participants
Started | 101 (Participant could enter follow up period even if the treatment period was not completed.) | 51
Completed | 101 | 50
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Daclatasvir + Sofosbuvir in Treatment-experienced Participants: Participants infected with hepatitis C virus (HCV) genotype-3 and previously exposed to an interferon formulation or sofosbuvir /ribavirin or any other anti-HCV agents therapy, received daclatasvir 60-mg and sofosbuvir 400-mg tablets orally once daily for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Daclatasvir + Sofosbuvir in Treatment-naive Participants | Daclatasvir + Sofosbuvir in Treatment-experienced Participants | Total
Number analyzed (Participants) | 101 | 51 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (10.73) | 56.3 (6.64) | 52.3 (9.94)
Age, Customized [Number; unit: participants]
  <65 years | 95 | 47 | 142
  >= 65 years | 6 | 4 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 19 | 62
  Male | 58 | 32 | 90

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Treatment-Naive Participants With Sustained Virologic Response at Follow-up Week 12 (SVR12) Target Detected (TD) or Target Not Detected (TND)
Description: SVR12 was defined as hepatitis C virus (HCV) RNA less than the lower limit of quantitation ie., 25 IU/mL, TD or TND at follow-up Week 12. HCV RNA levels were measured by the Roche Cobas® TaqMan® HCV Test version 2.0 from the central laboratory.
Time Frame: Week 12 (Follow-up period)
Population: The analysis was performed in all treated participants who received at least 1 dose of active study therapy.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Daclatasvir + Sofosbuvir in Treatment-naive Participants
Number analyzed (Participants) | 101
Percentage of participants | 90.1 [82.5 to 95.1]

2. Secondary Outcome: Percentage of Participants With Rapid Virologic Response at Week 4 (RVR) Target Not Detected (TND)
Description: RVR was defined as hepatitis C virus RNA levels to be < lower limit of quantitation ie, 25 IU/mL TND at Week 4. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory.
Time Frame: Week 4
Population: The analysis was performed in all treated participants who received at least 1 dose of active study therapy.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Daclatasvir + Sofosbuvir in Treatment-naive Participants | Daclatasvir + Sofosbuvir in Treatment-experienced Participants
Number analyzed (Participants) | 101 | 51
Percentage of participants | 63.4 [53.2 to 72.7] | 72.5 [58.3 to 84.1]

3. Secondary Outcome: Percentage of Participants With Complete Early Virologic Response (cEVR) Target Not Detected (TND)
Description: cEVR was defined as hepatitis C virus RNA levels to be < lower limit of quantitation ie, 25 IU/mL TND at Week 12. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory.
Time Frame: Week 12
Population: The analysis was performed in all treated participants who received at least 1 dose of active study therapy.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Daclatasvir + Sofosbuvir in Treatment-naive Participants | Daclatasvir + Sofosbuvir in Treatment-experienced Participants
Number analyzed (Participants) | 101 | 51
Percentage of participants | 98.0 [93.0 to 99.8] | 100.0 [93.0 to 100.0]

4. Secondary Outcome: Percentage of Participants With End of Treatment Response (EOTR) Target Not Detected (TND)
Description: EOTR were defined as hepatitis C virus RNA levels to be < lower limit of quantitation ie, 25 IU/mL TND at end of treatment. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory.
Time Frame: Up to the end of treatment (up to 24 weeks)
Population: The analysis was performed in all treated participants who received at least 1 dose of active study therapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Daclatasvir + Sofosbuvir in Treatment-experienced Participants: Participants infected with HCV genotype-3 and previously exposed to an interferon formulation or sofosbuvir /ribavirin or any other anti-HCV agents therapy, received daclatasvir 60-mg tablets and sofosbuvir 400-mg tablets orally once daily for 12 weeks.
Arm/Group | Daclatasvir + Sofosbuvir in Treatment-naive Participants | Daclatasvir + Sofosbuvir in Treatment-experienced Participants
Number analyzed (Participants) | 101 | 51
percentage of participants | 99.0 [94.6 to 100.0] | 100.0 [93.0 to 100.0]

5. Secondary Outcome: Percentage of Participants Who Achieved Hepatitis C Virus (HCV) RNA Levels Less Than the Lower Limit of Quantitation (LLOQ) - Target Not Detected (TND)
Description: Percentage of participants who achieved HCV RNA <LLOQ, TND was determined (LLOQ: 25 IU/mL). HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory.
Time Frame: Week 1, 2, 6, 8 (treatment period)
Population: The analysis was performed in all treated participants who received at least 1 dose of active study therapy.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Daclatasvir + Sofosbuvir in Treatment-naive Participants | Daclatasvir + Sofosbuvir in Treatment-experienced Participants
Number analyzed (Participants) | 101 | 51
Percentage of participants
  Week 1 | 11.9 [6.3 to 19.8] | 2.0 [0.0 to 10.4]
  Week 2 | 34.7 [25.5 to 44.8] | 29.4 [17.5 to 43.8]
  Week 6 | 86.1 [77.8 to 92.2] | 90.2 [78.6 to 96.7]
  Week 8 | 95.0 [88.8 to 98.4] | 98.0 [89.6 to 100.0]

6. Secondary Outcome: Percentage of Participants Who Achieved Hepatitis C Virus (HCV) RNA Levels Less Than the Lower Limit of Quantitation (LLOQ)- Target Detected (TD) or Target Not Detected (TND)
Description: Percentage of participants who achieved HCV RNA <LLOQ,TD or TND was determined (LLOQ: 25 IU/mL). HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory.
Time Frame: Week 1, 2, 4, 6, 8, 12, End of treatment (treatment period), Week 4 (follow-up period), Week 24 (follow-up period)
Population: The analysis was performed in all treated participants who received at least 1 dose of active study therapy.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Daclatasvir + Sofosbuvir in Treatment-naive Participants | Daclatasvir + Sofosbuvir in Treatment-experienced Participants
Number analyzed (Participants) | 101 | 51
Percentage of participants
  Week 1 | 39.6 [30.0 to 49.8] | 23.5 [12.8 to 37.5]
  Week 2 | 77.2 [67.8 to 85.0] | 68.6 [54.1 to 80.9]
  Week 4 | 94.1 [87.5 to 97.8] | 98.0 [89.6 to 100.0]
  Week 6 | 100.0 [96.4 to 100.0] | 98.0 [89.6 to 100.0]
  Week 8 | 100.0 [96.4 to 100.0] | 100.0 [93.0 to 100.0]
  Week 12 | 98.0 [93.0 to 99.8] | 100.0 [93.0 to 100.0]
  End of treatment | 99.0 [94.6 to 100.0] | 100.0 [93.0 to 100.0]
  Follow-up Week 4 | 91.1 [83.8 to 95.8] | 86.3 [73.7 to 94.3]
  Follow-up Week 24 | 89.1 [81.3 to 94.4] | 82.4 [69.1 to 91.6]

7. Secondary Outcome: Percentage of Participants With Or Without Cirrhosis at Baseline Who Achieved Sustained Virologic Response at Follow-up Week 12 (SVR12)
Description: SVR12 was defined as hepatitis C virus (HCV) RNA less than the lower limit of quantitation ie. 25 IU/mL, target detected or target not detected at follow-up Week 12. Cirrhosis was considered a negative predictor of SVR in participants treated with an interferon formulation or ribavirin. Presence or absence of cirrhosis was determined at baseline and follow-up Week 12 in the participants to evaluate the post-treatment relapse.
Time Frame: Baseline, Week 12 (Follow-up period)
Population: The analysis was performed in all treated participants who received at least 1 dose of active study therapy. The 'n' signifies the number of evaluable participants with or without cirrhosis in the reporting arm and time point, respectively.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Daclatasvir + Sofosbuvir in Treatment-naive Participants | Daclatasvir + Sofosbuvir in Treatment-experienced Participants
Number analyzed (Participants) | 101 | 51
Percentage of participants
  With cirrhosis (n= 19, 13) | 57.9 [33.5 to 79.7] | 69.2 [38.6 to 90.9]
  Without cirrhosis (n= 75, 34) | 97.3 [90.7 to 99.7] | 94.1 [80.3 to 99.3]

8. Secondary Outcome: Percentage of Participants With CC or Non-CC Genotype at the IL28B rs12979860 Single Nucleotide Polymorphisms (SNPs) Who Achieved Sustained Virologic Response After 12 Weeks of Follow-up (SVR12)
Description: Participants categorized into 2 genotypes (CC and non-CC) based on SNPs in the IL28B gene were assessed for SVR12, defined as response in which hepatitis C virus (HCV) RNA levels below lower limit of quantitation (LLOQ) below target detected or target not detected at follow-up Week 12 (LLOQ: 25 IU/mL). HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory.
Time Frame: Week 12 (Follow-up period)
Population: The analysis was performed in all treated participants who received at least 1 dose of active study therapy. Here, ''n'' signifies number of participants evaluable for the specified category.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Daclatasvir + Sofosbuvir in Treatment-naive Participants | Daclatasvir + Sofosbuvir in Treatment-experienced Participants
Number analyzed (Participants) | 101 | 51
Percentage of participants
  Genotype: CC (n=40, 20) | 90.0 [76.3 to 97.2] | 95.0 [75.1 to 99.9]
  Genotype: Non-CC (n=61, 31) | 90.2 [79.8 to 96.3] | 80.6 [62.5 to 92.5]

9. Primary Outcome: Percentage of Treatment-Experienced Participants With Sustained Virologic Response at Follow-up Week 12 (SVR12) Target Detected (TD) or Target Not Detected (TND)
Description: SVR12 was defined as hepatitis C virus (HCV) RNA less than the lower limit of quantitation ie., 25 IU/mL, target detected or target not detected at follow-up Week 12. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory.
Time Frame: Week 12 (Follow-up period)
Population: The analysis was performed in all treated participants who received at least 1 dose of active study therapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Daclatasvir + Sofosbuvir in Treatment-experienced Participants: Participants infected with HCV genotype-3 and previously exposed to an interferon formulation or sofosbuvir /ribavirin or any other anti-HCV agents therapy, received daclatasvir 60-mg and sofosbuvir 400-mg tablets orally once daily for 12 weeks.
Arm/Group | Daclatasvir + Sofosbuvir in Treatment-experienced Participants
Number analyzed (Participants) | 51
percentage of participants | 86.3 [73.7 to 94.3]

10. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Discontinuations Due to Adverse Events (AEs)
Description: AE was defined as any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that does not necessarily have a causal relationship with treatment. SAE was defined as a medical event that at any dose resulted in death, persistent or significant disability/incapacity, or drug dependency/abuse; was life-threatening, an important medical event, or a congenital anomaly/birth defect; or required or prolonged hospitalization.
Time Frame: From Day 1 first dose to last dose plus 7 days
Population: The analysis was performed in all treated participants who received at least 1 dose of active study therapy.
Measure: Number; unit: Participants
Arm/Group | Daclatasvir + Sofosbuvir in Treatment-naive Participants | Daclatasvir + Sofosbuvir in Treatment-experienced Participants
Number analyzed (Participants) | 101 | 51
Participants
  SAEs | 1 | 0
  Discontinuations Due to AEs | 0 | 0

ADVERSE EVENTS:
Time Frame: From Day 1 first dose to last dose plus 7 days
Description: On-treatment period.
Groups:
- Daclatasvir + Sofosbuvir: All participants infected with hepatitis C virus (HCV) genotype-3 received daclatasvir 60-mg tablets and sofosbuvir 400-mg tablets orally once daily for 12 weeks during the study.
Arm/Group | Daclatasvir + Sofosbuvir
Serious Adverse Events (participants affected / at risk) | 1/152
Other Adverse Events (participants affected / at risk) | 73/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Daclatasvir + Sofosbuvir (N=152)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Daclatasvir + Sofosbuvir (N=152)
Abdominal pain (Gastrointestinal disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 13
Fatigue (General disorders) | 29
Headache (Nervous system disorders) | 30
Insomnia (Psychiatric disorders) | 9
Nausea (Gastrointestinal disorders) | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.